CLINICAL TRIAL: NCT01413802
Title: Intra Operative Continuous Laryngeal Nerve Monitoring During Thyroid Surgery and Interpretation of the Post-operative Voice Quality in Relation to the Electromyography Data Obtained During Surgery
Acronym: CoNeMoTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011/371
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Thyroid Surgery
Keywords: Thyroid surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thyroid surgery. (Experimental): Patients who undergo thyroid surgery during which intra operative continuous nerve monitoring will be used.
  Interventions: Procedure: Continuous nerve monitoring

INTERVENTIONS:
Procedure: Continuous nerve monitoring — Continuous nerve monitoring is performed during thyroid surgery.

SUMMARY:
During thyroid surgery the laryngeal recurrent nerves (and for this reason the voice quality) are at risk. Therefore intra operative continuous neuromonitoring could help to prevent harm to these nerves. Electromyographic data (EMG values) are collected during surgery (1). In the postoperative follow-up period detailed voice analysis is performed (2): subjective auditive perceptive evaluation and videostroboscopy. Analysis and comparison of (1) and (2) will be performed in order to find out if we can find a predictive correlation between the EMG data (1) and the voice quality (2).

ELIGIBILITY:
Inclusion Criteria:

* patients (men/women) requiring thyroid surgery

Exclusion Criteria:

* patients younger than 18 years, patients with preoperative vocal cord anatomical and functional anomalies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2012-02-28 (Actual); Study Completion 2013-03-05 (Actual)

PRIMARY OUTCOMES:
Detailed voice analysis to find a predictive correlation between the EMG data and the voice quality, after thyroid surgery. | 1 week after surgery
  The primary outcome is to check if by continuous vagal nerve stimulation reversible damage to the recurrent laryngeal nerve can be foreseen, and therefore avoided. The detailed voice analysis that is used, consist of subjective auditive perceptive evaluation and videostroboscopy.
Detailed voice analysis to find a predictive correlation between the EMG data and the voice quality, after thyroid surgery. | 3 weeks after surgery
  The primary outcome is to check if by continuous vagal nerve stimulation reversible damage to the recurrent laryngeal nerve can be foreseen, and therefore avoided. The detailed voice analysis that is used, consist of subjective auditive perceptive evaluation and videostroboscopy.
Detailed voice analysis to find a predictive correlation between the EMG data and the voice quality, after thyroid surgery. | 3 months after surgery
  The primary outcome is to check if by continuous vagal nerve stimulation reversible damage to the recurrent laryngeal nerve can be foreseen, and therefore avoided. The detailed voice analysis that is used, consist of subjective auditive perceptive evaluation and videostroboscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Vermeersch, MD Phd, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Onze Lieve Vrouw clinic Aalst, Aalst
  - University Hospital Ghent, Ghent

REFERENCES:
- See also: Related Info — http://www.uzgent.be